CLINICAL TRIAL: NCT01312259
Title: Clinical Efficacy of Changing the InterStim® Parameters in Patients With Interstitial Cystitis/Painful Bladder Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pelvic and Sexual Health Institute (Other)
Responsible Party: Principal Investigator, Kristene Whitmore, M.D., Medical Director, Pelvic and Sexual Health Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 19522
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Painful Bladder Syndrome; Interstitial Cystitis; Pelvic Floor; Insufficiency; Bowel Dysfunction; Sexual Dysfunction; Pelvic Floor; Incompetency
Keywords: Painful Bladder Syndrome; Interstitial Cystitis; Pelvic Floor dysfunction; Fecal incontinence; Constipation; Sexual dysfunction; Dyspareunia; Vulvodynia
MeSH Terms: conditions — Cystitis, Interstitial; Intestinal Diseases; Sexual Dysfunction, Physiological; Fecal Incontinence; Constipation; Dyspareunia; Vulvodynia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interstim Parameter Frequency 14 HZ (Active Comparator): Subjects in this arm will receive 14 Hx as their frequency for the first three months. For the second 3 months, these patients will receive 40 Hz. Six months after the devise has been implanted, the patient has the option to choose which frequency they feel allows for better symptom control, and this is how the devise will be programmed.
  Interventions: Other: Changing the Interstim parameter of '' Frequency" in patients with Interstitial Cystitis
- Interstim Parameter Frequency 40 HZ (Experimental): Subjects in this arm will receive 40 Hz as their frequency for the first three months. For the second 3 months, these patients will receive 14 Hz. Six months after the devise has been implanted, the patient has the option to choose which frequency they feel allows for better symptom control, and this is how the devise will be programmed.
  Interventions: Other: Changing the Interstim parameter of '' Frequency" in patients with Interstitial Cystitis

INTERVENTIONS:
Other: Changing the Interstim parameter of '' Frequency" in patients with Interstitial Cystitis — Subjects will be randomized into one of two groups. Group One will be programmed to receive 14 Hz as their frequency, while the other group (Group 2) will receive 40 Hz as their frequency for the first ninety days after surgical implantation. After three months each patient will come in to the office to have their InterStim frequency changed to the opposite frequency. After each patient has had three months to evaluate each of the two frequencies, the next step is to allow the patient to decide which setting they thought best controlled their respective symptoms. The InterStim was then programed to whichever frequency the patient chose, and this would remain for three to six months.
  Other Names: InterStim; Sacralneuromodulation device; IPG (Implantable pulse generator)

SUMMARY:
Purpose:

1. To demonstrate better symptoms control (pain, urinary urgency and frequency) with sacral neuromodulation (SNM) in patients with interstitial cystitis /painful bladder syndrome (IC/PBS) using a stimulation frequency of 40 hertz (experimental) compared to a frequency of 14 hertz (standard).
2. The evaluate the efficacy of the two frequency settings on the other associated conditions that often coexist in patients with IC/PBS, such as female sexual dysfunction (FSD), bowel dysfunction, high tone pelvic floor dysfunction (HTPFD, painful spasm of the pelvic floor muscles), Vulvodynia (pain at the opening of the vagina).

DETAILED DESCRIPTION:
Purpose:

1. Primary: to demonstrate better symptoms control (pain, urinary urgency and frequency) with sacral neuromodulation (SNM) in patients with interstitial cystitis /painful bladder syndrome (IC/PBS) using a stimulation frequency of 40 hertz (experimental) compared to a frequency of 14 hertz (standard).
2. Secondary: The evaluate the efficacy of the two frequency settings on the other associated conditions that often coexist in patients with IC/PBS, such as female sexual dysfunction (FSD), bowel dysfunction, high tone pelvic floor dysfunction (HTPFD, painful spasm of the pelvic floor muscles), Vulvodynia (pain at the opening of the vagina).

ELIGIBILITY:
Inclusion Criteria:

* Female with diagnosis of IC/PBS with implanted IPG Interstim.
* Scores > 8 on the Interstitial Cystitis Symptom index questionnaire (ICSI) and > 8 on the Interstitial Cystitis Problem Index questionnaire (ICPI).
* Signed Informed Consent.

Exclusion Criteria:

* Progressive neurologic disease or peripheral neuropathy.
* History of bladder surgery.
* Subjects implanted with other neuromodulation device.
* Current or planning pregnancy; Breastfeeding.
* Subjects who are not deemed able to fill questionnaires
* Mental illness or mentally unstable patients

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2011-04; Primary Completion 2017-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Improvement in Urinary symptoms and Bladder pain/discomfort | 1 year
  To demonstrate better symptoms control (pain, urinary urgency and frequency) with sacral neuromodulation (SNM) in patients with interstitial cystitis /painful bladder syndrome (IC/PBS) using a stimulation frequency of 40 hertz (experimental) compared to a frequency of 14 hertz (standard).

SECONDARY OUTCOMES:
Improvement in Bowel symptoms and Sexual Function | 1 year
  The evaluate the efficacy of the two frequency settings on the other associated conditions that often coexist in patients with IC/PBS, such as female sexual dysfunction (FSD), bowel dysfunction, high tone pelvic floor dysfunction (HTPFD, painful spasm of the pelvic floor muscles), Vulvodynia (pain at the opening of the vagina).

CONTACTS AND LOCATIONS:
Overall Officials: Kristene E Whitmore, MD, Principal Investigator — Drexel University College of Medicine
Locations (1):
- Pelvic and Sexual Health Institute, Philadelphia, Pennsylvania, United States